CLINICAL TRIAL: NCT04499326
Title: Use of Patient Reported Outcome Measures (PROMs) to Assess Quality of Life and Economic Evaluation of Cardiac Catheter Ablation of Ventricular Tachycardia: a Feasibility and Cohort Study
Brief Title: Improving Patient Reported Outcome Measures in Catheter Ablation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: University College, London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRAS 264743
Record Dates: First submitted 2020-07-31; First posted 2020-08-05 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Ventricular Tachycardia; ICD; Quality of Life
Keywords: Catheter ablation; Patient reported outcome measure; Incremental cost effectiveness ratio
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients undergoing catheter ablation of VT
  Interventions: Other: Validated quality of life questionnaire (EQ-5D & C-CAP)
- Comparator (Active Comparator): Patients undergoing AAD therapy for VT
  Interventions: Other: Validated quality of life questionnaire (EQ-5D & C-CAP)

INTERVENTIONS:
Other: Validated quality of life questionnaire (EQ-5D & C-CAP) — Patient quality of life to be assessed at baseline, 1, 2, 3, 4, 6, 9 and 12 months

SUMMARY:
This study will assess whether more frequent measurement of patient reported outcome measures (PROMs) - specifically health related quality of life (HRQL) - can improve the evaluation of the clinical effectiveness and cost-effectiveness of catheter ablation of ventricular tachycardia (VT) in patients with an Implantable Cardioverter Defibrillator (ICD).

It is designed to have feasibility outcomes which contribute to answering the above.

DETAILED DESCRIPTION:
Patients who have been implanted with an ICD are at risk of suffering from dangerous arrhythmias such as VT.

Patients can experience clinical events including worsening of any underlying heart failure regardless of either VT ablation or medical therapy treatment strategy (anti-arrhythmic drugs (AAD)). VT ablation is a specialist procedure which has been proven in randomised clinical trials (RCTs) to confer symptomatic relief from VT, reduced hospitalisations and reduced shocks from ICDs. However, there is no effect on mortality.

The frequent nature of clinical events in this group of patients may affect their health status quite dramatically and yet based on current trial evidence, only 3 out of 6 randomised trials in VT ablation reported PROMs. This can lead to brittle conclusions about the overall cost-effectiveness profile of a procedure such as VT ablation.

This study will assess for the feasibility of more frequent HRQL monitoring and its impact on whether it is able to better capture the clinical narrative and quality of life changes of patients with severe heart failure and an ICD. And thus the assessment of both clinical effectiveness and cost effectiveness of catheter ablation of VT or continuing anti arrhythmic drug therapy.

METHOD & SETTING Single centre study at St Bartholomew's Hospital London. Patients will be identified through established local pathways - there are traditional outpatient specialist clinics where Consultant Cardiologists receive referrals of patients for consideration of managing patients with VT, including ablation. In addition, there are joint VT clinics operated by Consultants as well as by cardiac physiologists. In the outpatient VT clinic, 85 patients were seen in a 10-month window - it is assumed that this scale will allow feasible identification of patients to be recruited to the both the groups of this study.

ELIGIBILITY:
Inclusion Criteria:

Adults (>18 years) With an Implantable Cardioverter Defibrillator (ICD) implanted >3 months from time of recruitment and a previous episode of documented VT requiring therapy from the ICD.

And impaired LV/RV function Willing and able to give written informed consent

Exclusion Criteria:

Patients who are planning to move away from study site within 12 months of enrolment who wished to use postal method to complete their HRQL Patients who are unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Completion rate of HRQL forms for patients undergoing VT ablation and those starting or continuing AAD therapy | 1 year follow up

SECONDARY OUTCOMES:
Recruitment rate of patients who fulfil study criteria | 1 year
- Patient preferences for either paper or electronic HQRL (as a percentage of total recruitment) | 1 year
Patient reported HRQL of VT ablation and AAD therapy on both EQ-5D and C-CAP | 18 months
Impact on the cost-effectiveness calculation of VT ablation (using EQ-5D, and a number of different EQ-5D data points) | 18 months
  Using the Incremental Cost-effectiveness ratio

CONTACTS AND LOCATIONS:
Overall Officials: Pier Lambiase, PhD, Study Chair — UCL
Locations (1):
- St Bartholomew's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for outcome measures will be made available
Supporting Information: CSR
Time Frame: In accordance with NHS Research governance framework
Access Criteria: Upon reasonable request